CLINICAL TRIAL: NCT06071390
Title: The Effect of Animation-Assisted Information Video Viewing on Fear and Anxiety in Children Before Endoscopy Procedure: A Randomized Controlled Study
Brief Title: The Effect of Animation-Assisted Information Video Viewing on Fear and Anxiety in Children Before Endoscopy Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Merve Koyun, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Endoscopy
Record Dates: First submitted 2023-09-27; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Endoscopy; Animation; Fear; Anxiety; Child
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled experimental study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children watching animated- assisted video before endoscopy procedure (Experimental): Inclusion criteria were children and mothers who voluntarily participated, who were aged 6-12 years, who know Turkish, and who do not have a vision or mental problem at a level to watch the image.
  Interventions: Behavioral: Animated- assisted video
- Children not watching animated- assisted video before endoscopy procedure (No Intervention): Exclusion criteria were children and mothers who not voluntarily participated, who were not aged 6-12 years, who don't know Turkish, and who have a vision or mental problem at a level to watch the image.

INTERVENTIONS:
Behavioral: Animated- assisted video — For the experimental group, 15 minutes prior to the endoscopy, the researcher provided insight into the procedure by showing them a 3-minute animated video titled "Endocan." This video, crafted by Köse in 2019 for his doctoral dissertation, offers a succinct overview of the endoscopy procedure.
  Arms: Children watching animated- assisted video before endoscopy procedure

SUMMARY:
The aim of this study was to evaluate watching video about procedure on reduce anxiety and fear in children before the endoscopy.

DETAILED DESCRIPTION:
Being admitted to a hospital is an inherently stressful event for both children and their parents, regardless of the reason In such a context where children experience multifaceted effects, it becomes imperative to ensure that their hospital experience is as positive as possible. Hospitalized children often undergo medical procedures such as blood sampling, venipuncture, invasive drug administration, lumbar puncture, and intrathecal drug administration. These interventions, whether diagnostic or therapeutic, are sources of fear and anxiety for them. With a surge in gastrointestinal system disorders in children, the use of endoscopy, both as a diagnostic and therapeutic tool, has become more prevalent. Pediatric nurses play a pivotal role in alleviating the fear and anxiety experienced by children and their families during medical procedures, ensuring a smoother adjustment to the process. Prior research indicates that children's fear and anxiety levels significantly decrease, and parental satisfaction rises when children are informed about impending medical procedures. Moreover, providing pre-procedure information has been linked to heightened treatment compliance, expedited recovery post-procedure, and a reduced reliance on analgesics. While tailored educational programs are highly effective in conveying information about medical procedures or diseases to children, their elevated cost restricts widespread implementation. Traditional, cost-effective teaching strategies such as oral presentations, brochures, and booklets, although tailored for school-age children, haven't demonstrated consistent efficacy in enhancing clinical results. It has been noted that insufficient information provision can make children reliant on parents for clarification, with most procedural details tailored to parental understanding. In response, evidence-based initiatives have been introduced to enhance educational quality, boost patient clinical outcomes, and ensure cost-effectiveness. Given children's developmental stage, diverse educational techniques have been employed to prepare them for medical procedures, including endoscopy. An emerging method involves utilizing cartoons, which, when effectively employed, blend entertainment with instruction.

ELIGIBILITY:
Inclusion Criteria:

* Children and mothers who voluntarily participated,
* who were aged 6-12 years,
* who know Turkish,
* who do not have a vision or mental problem at a level to watch the image.

Exclusion Criteria:

* children and mothers who not voluntarily participated,
* who were not aged 6-12 years,
* who don't know Turkish,
* who have a vision or mental problem at a level to watch the image.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
changing the anxiety | 'Before watching video' and 'After watching video, within 5 minutes'
  Children's Anxiety Meter- State (CAM-S) is designed like a thermometer, featuring a bulb at its base and horizontal markers at regular intervals as it ascends. Children are asked to represent their feelings on this scale by marking where they stand "right now". They are instructed, "Imagine that all your anxious or angry feelings are on the bulb or bottom part of the thermometer. If you are a little worried or nervous, the feelings may go up a little on the thermometer. If you are very, very anxious or nervous, emotions can go all the way to the top. Put a line on the thermometer showing how anxious or nervous you are." This scale provides scores ranging from 0 to 10. As the score increases, the level of anxiety increases.
changing the fear | 'Before watching video' and 'After Watching Video, within 5 minutes'
  The Children's Fear Scale (CFS) was developed by Chambers et al. in 2011. It was adapted into Turkish by Gerceker et al. in 2018. It comprises five facial expressions ranging from neutral to extreme fear. Both researchers and family members can use the CFS to measure fear and anxiety in children before and during procedures. This scale provides scores ranging from 0-4. As the score increases, the level of fear increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
other researchers may view the study once it is published.

REFERENCES:
- [Background] Alvarez-Garcia C, Yaban ZS. The effects of preoperative guided imagery interventions on preoperative anxiety and postoperative pain: A meta-analysis. Complement Ther Clin Pract. 2020 Feb;38:101077. doi: 10.1016/j.ctcp.2019.101077. Epub 2019 Dec 4. PMID 32056813
- [Background] Arican, Ş., Yücel, A., Yılmaz, R., Hacıbeyoğlu, G., Yusifov, M., Yüce, S., Topal, A.(2020). Anxiety level and risk factors among pediatric patients in endoscopic procedures outside the operating room: A cross-sectional study. J Surg Med, 4(8), 693-697.
- [Background] Camur Z, Sarikaya Karabudak S. The effect of parental participation in the care of hospitalized children on parent satisfaction and parent and child anxiety: Randomized controlled trial. Int J Nurs Pract. 2021 Oct;27(5):e12910. doi: 10.1111/ijn.12910. Epub 2020 Dec 16. PMID 33331038